CLINICAL TRIAL: NCT06322238
Title: A Multi-gene Pharmacogenetic Panel to Prevent Adverse Drug Reactions in Daily Primary Care Practice: Open-label, Mayo Clinic Multisite (Mayo Clinic Health System-Rochester Primary Care), Controlled, Implementation Study Taking the Results of the PREPARE Study Into Minnesota (PREPARE-Mayo)
Brief Title: Pharmacogenetic Panel to Prevent Adverse Drug Reactions in Daily Primary Care Practice:
Acronym: PREPARE-Mayo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Isa J. Houwink, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-008706
Record Dates: First submitted 2024-02-09; First posted 2024-03-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pharmacogenomic Drug Interaction; Side Effect of Drug; Ineffective Drug Action; Drug Metabolism, Poor, CYP2D6-Related; Drug Metabolism, Poor, CYP2C19-Related
Keywords: pharmacogenomics; PGx; CPIC; primary care; drug metabolism; side effects; ineffectiveness; PREPARE-Mayo
MeSH Terms: conditions — Drug Metabolism, Poor, CYP2D6-Related; Drug Metabolism, Poor, CYP2C19-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGx testing arm (Experimental)
  Interventions: Diagnostic Test: PGx panel test
- Delayed PGx testing arm (Placebo Comparator)
  Interventions: Diagnostic Test: PGx panel test

INTERVENTIONS:
Diagnostic Test: PGx panel test — In this prospective, non-randomized, step-wedge design controlled clinical study (PREPARE-MAYO Rochester, Mayo Clinic Health System), pre-emptive genotyping of a panel of clinically relevant PGx-markers, for which CPIC guidelines are available.

SUMMARY:
The purpose of this study is to determine whether the implementation of pre-emptive pharmacogenomic (PGx) testing of a panel of clinically relevant PGx markers, to guide the dose and drug selection for 39 commonly prescribed drugs, will result in an overall reduction in the number of clinically relevant drug-genotype associated ADRs which are causally related to the initial drug of inclusion (referred to as 'index drug').

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject must be ≥ 18 years old
2. Subject must receive a 1st prescription (meaning no known prescription for this drug in the preceding 12 months) for a drug included in Table 1, which is prescribed to them in routine primary care.
3. Subject is able and willing to take part and willing to be followed up on for 48 weeks
4. Subject is able to donate saliva
5. Subject has signed informed consent
6. Subject meets requirement for computer access implying computer literacy as measured by active use of the patient portal or their email

Exclusion Criteria:

1. For the investigational arm only: Previous (direct-to-consumer, or clinical) pharmacogenomic testing that includes any of the genes included in the Focused Pharmacogenomics Panel
2. Pregnant or lactating (to be verbally confirmed with the patient)
3. Life expectancy estimated to be less than three months as determined by patient receiving hospice care
4. Duration of index drug total treatment length is planned to be less than seven consecutive days.
5. Current inpatients
6. Unable to consent to the study
7. Unwilling to take part
8. Subject has no permanent address
9. Subject has no current primary care provider
10. Subject is, in the opinion of the study coordinator after discussion with participating clinician/pharmacist/investigator, not suitable to participate in the study
11. Patient has a diagnosis of stage 4 or 5 chronic kidney disease (CKD) or is receiving dialysis
12. Patients with advanced liver failure (stage Child-Pugh C) or a diagnosis of liver cirrhosis
13. History of a liver transplant or an allogeneic hematopoietic stem cell transplant
14. DNA sample collected that requires retesting in the event that DNA collected was not sufficient for testing as determined by the laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Drug Reaction (ADR) | 48 weeks
  The count of participants who experience any of the following ADR's: muscle aches, falling, tripping, fainting, palpations, emotional changes, or physical changes

SECONDARY OUTCOMES:
PREPARE-MAYO Clinicians' and pharmacists' Questionnaire. | 48 weeks
  The 29-item PREPARE-MAYO Clinicians' and pharmacists' Questionnaire measures the Experience and Attitude, Knowledge, Knowledge testing and Needs assessment of clinicians and pharmacists. Each item is scored from 1 (disagree) to 4 (agree). Total possible scores range from 29 to 116, with lower scores indicating less knowledge and higher scores indicating more knowledge.
Patient-Reported Outcomes Measurement Information System (PROMIS-10) Global Health Questionnaire | 48 weeks
  The 10-item PROMIS Global Health measures general, physical, mental and social health. Each item is scored from 1 (poor health) to 5 (excellent health). Total possible scores range from 10 to 50, with lower scores indicating worse state of health and higher scores indicating greater state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Isa Houwink, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginniing 9 to 36 months following publication provided the investigator who proposes the use of the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data sharing use /sharing agreement with Mayo Clinic and the PI.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials